CLINICAL TRIAL: NCT03415646
Title: The Effect of Double Injection Erector Spinae Plane Block on Postoperative Pain Following Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Can AKSU, Assistant Professor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2017-377
Record Dates: First submitted 2018-01-10; First posted 2018-01-30 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Postoperative Pain; Breast Cancer
Keywords: erector spinae plane block; breast surgery; postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block Group (Active Comparator): Erector Spinae Plane Block administered group
  Interventions: Other: Erector Spinae Plane Block; Device: Intravenous Morphine patient controlled analgesia device
- Control Group (Sham Comparator): Control group
  Interventions: Device: Intravenous Morphine patient controlled analgesia device

INTERVENTIONS:
Other: Erector Spinae Plane Block — erector spinae plane block with double level injection will be administered before the surgery
  Arms: Block Group
Device: Intravenous Morphine patient controlled analgesia device — 24 hour morphine consumption will be recorded

SUMMARY:
Postoperative analgesia in breast surgery is a difficult and overworked issue due to extensive surgery and complex innervation of the breast. Erector spinae plane block (ESB) is a new defined regional anesthesia technique for thoracic analgesia.Main purpose of this study was to evaluate the analgesic effect of ultrasound guided double injection ESB in breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* 25-70 years of age
* ASA I-II
* Undergoing elective breast cancer surgery

Exclusion Criteria:

* obesity (body mass index >35 kg/m2)
* infection of the skin at the site of needle puncture area
* patients with known allergies to any of the study drugs
* coagulopathy
* recent use of analgesic drugs.

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-02-03 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | 24 hour postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University Hospital, İzmit, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No